CLINICAL TRIAL: NCT03489109
Title: 2-5 Intermittent Caloric Restriction for Weight Loss and Insulin Resistance in HIV-Infected Adults With Features of the Metabolic Syndrome
Brief Title: 2-5 Intermittent Caloric Restriction in HIV
Acronym: 2-5toWIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow/Insufficient accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180075
Record Dates: First submitted 2018-04-04; First posted 2018-04-05 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2021-12

CONDITIONS: Human Immunodeficiency Virus; Metabolic Syndrome
Keywords: Fasting
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Metabolic Syndrome; Fasting | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting diet (Experimental): HIV positive subjects with body mass index ≥30 kg/m2 (obese) consume approximately 25% of their daily calories for 2 non-consecutive days per week, normal diet for the other 5 days, and receive healthy lifestyle counseling for 12 weeks.
  Interventions: Behavioral: Intermittent fasting
- Standard of Care diet (Active Comparator): HIV positive subjects with body mass index ≥30 kg/m2 (obese) receive nutritional and healthy lifestyle counseling for 12 weeks.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Intermittent fasting — Subject will consume approximately 25% of their daily calories for 2 days per week. The other 5 days they will eat their normal diet
  Arms: Intermittent Fasting diet
Other: Standard of Care — Subject will receive standard of care recommendations for healthy diet and lifestyle
  Arms: Standard of Care diet

SUMMARY:
Background:

Weight gain can lead to obesity and diabetes even in people living with human immunodeficiency virus (HIV). Researchers want to see if the technique intermittent calorie restriction can help overweight people with HIV as an alternative to traditional diets.

Objective:

To see if intermittent calorie restriction leads to weight loss and improved blood sugar in obese people with HIV.

Eligibility:

Adults ages 18-65 with HIV who are obese and do not have diabetes

Design:

Participants will be screened with a medical history, physical exam, and blood and urine tests.

Before starting treatment, participants will:

* Have a nutritional consultation
* Get a pedometer to record daily steps
* Test a restricted diet for 1 day
* Have a body x-ray

At the baseline visit, participants will have:

* Blood drawn after they drink a sugar drink
* Questions about their health and eating
* A nutritional consultation
* Resting energy expenditure measured. Participants will fast overnight. Then they will lie down while a plastic bubble goes over the head and a plastic sheet covers the upper body. Oxygen flows into the bubble.
* Liver stiffness test. A wand on the stomach releases sound waves like an ultrasound.

For 12 weeks, some participants will be on a standard diet. Others will restrict how much food they eat 2 days a week. On those days they will eat about 25% of their recommended calories.

Participants will keep a diary of their diet and steps.

Participants will have 4 visits during the 12-week diet and 1 visit 12 weeks after the diet ends. They will repeat previous tests.

DETAILED DESCRIPTION:
The high prevalence of obesity coupled with chronic inflammation and immune activation places human immunodeficiency virus (HIV)-infected individuals at increased risk for metabolic complications emphasizing the need for more aggressive management of obesity and related co-morbidities in the aging HIV-infected population. The most effective treatment for obesity and metabolic syndrome is lifestyle modification, usually with a combination of caloric restriction and increased exercise. Intermittent caloric restriction (ICR) or intermittent fasting simplifies caloric restriction by severely limiting calories only a few days per week and allowing ad lib diet on the other days. Weight loss benefits are similar to those seen with conventional diets, however, data suggests possible added health benefits from intermittent fasting.

We propose to study the benefits of a 2-5 ICR strategy on weight, insulin resistance, and cardiovascular disease markers in obese HIV-infected adults with features of the metabolic syndrome. In a prospective pilot study, 50 HIVinfected adults will be randomized 1:1 to ICR or standard-of-care instruction of healthy diet and lifestyle for a 12-week intervention period. We hypothesize that ICR (2 days per week) will be an effective and acceptable diet strategy that will result in significant weight reduction, improvements in insulin sensitivity, and related metabolic parameters.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Aged 18 to 65 years
2. HIV RNA level less than or equal to 200 copies/mL for greater than or equal to1 year (1 measure greater than or equal to 200 allowed if also <500 and preceded and followed by one or more undetectable values)
3. Cluster of differentiation 4 (CD4) >200 cells/mL and no active opportunistic infection or malignancy
4. BMI greater than or equal to 30 kg/m^2
5. One or more components of the metabolic syndrome as defined below.

   * Risk Factor: Waist circumference

     * Men: Defining Level: >102 cm
     * Women: Defining Level: >88 cm
   * Risk Factor: Triglycerides, greater than or equal to 150 mg/dL
   * Risk Factor: High density lipoprotein (HDL) cholesterol

     * Men: Defining Level: <40 mg/dL
     * Women: Defining Level: <50 mg/dL
   * Risk Factor: Blood pressure, greater than or equal to 130 / greater than or equal to 85 mmHg
   * Risk Factor: Fasting glucose, greater than or equal to 110 mg/dL
6. Fasting blood glucose >60 mg/dL at screening
7. Willingness to allow sample storage for future research
8. Able to provide informed consent

EXCLUSION CRITERIA:

1. Established diagnosis of diabetes mellitus use of anti-diabetes medications, or a hemoglobin A1C (HgbA1C) of >7.0%
2. History of eating disorder, uncontrolled mood or thought disorder, significant gastrointestinal disorder or malabsorption, or significant hepatic or renal impairment
3. Current use of medical therapy for overweight/obesity including phentermine, orlistat, lorcaserin, naltrexone/bupropion, and liraglutide or history of weight loss surgery. Concomitant use of medications with side effects known to potentially influence appetite are allowed if on a stable dose for at least 12 months
4. History of symptomatic hypoglycemia.
5. Use of systemic glucocorticoids (stable dose daily inhaled corticosteroid allowed)
6. Chronic viral hepatitis C; subjects with a history of hepatitis C successfully treated can enroll >12 months after sustained virologic response
7. Alcohol or substance use disorder in the past year as defined by Diagnostic and Statistical Manual (DSM)-V or positive urine drug screen
8. Current pregnancy, actively seeking to become pregnant or breastfeeding
9. Any serious health or other condition which, in the opinion of the PI or their designee, could potentially interfere with the ability of a subject to comply with the procedures and assessments of the protocol or to safely participate and complete the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Hadigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-I-0075.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 35 subjects who were consented to protocol, four subjects withdrew prior to start of study, one subject was screen failure and 30 subjects started the study.
Groups:
- Intermittent Fasting Diet: HIV positive subjects with body mass index =30 kg/m2 (obese) consume approximately 25% of their daily calories for 2 non-consecutive days per week, normal diet for the other 5 days, and receive healthy lifestyle counseling for 12 weeks.
- Standard of Care Diet: HIV positive subjects with body mass index =30 kg/m2 (obese) receive nutritional and healthy lifestyle counseling for 12 weeks.
Period: Overall Study
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Started | 14 | 16
Completed | 13 | 14
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 10 | 14 | 24
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 2 | 3 | 5
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: kilograms] | 112.1 (18.4) | 109.6 (14.9) | 110.8 (16.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: The effect of intermittent fasting was measured by change in weight between baseline and at week 12
Time Frame: Assessed before 12-week intervention (baseline) and at week 12
Population: Analysis only includes subjects who completed through Week 12
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Intermittent Fasting Diet: Persons living with HIV and with body mass index >/= 30 kg/m2 (obese) consume approximately 25% of their daily calories for 2 non-consecutive days per week, normal diet for the other 5 days, and receive healthy lifestyle counseling for 12 weeks.
- Standard of Care Diet: Persons living with HIV and with body mass index >/= 30 kg/m2 (obese) receive nutritional and healthy lifestyle counseling for 12 weeks.
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Number analyzed (Participants) | 14 | 15
kilograms | -1.5 (4.9) | -1.8 (3.8)

2. Primary Outcome: Change in Insulin Sensitivity
Description: The effect of intermittent fasting on insulin sensitivity was measured by change in homeostatic model assessment of insulin resistance (HOMA-IR) between baseline and week 12. Homeostasis model assessment of insulin resistance (HOMA-IR) is a method to measure insulin sensitivity. Optimal insulin sensitivity is a HOMA-IR ratio less than 1. Levels above 1.9 signal early insulin resistance, while levels above 2.9 signal significant insulin resistance.
Time Frame: Assessed before 12-week intervention (baseline) and at week 12
Population: Analysis only includes subjects who completed study through Week 12
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Number analyzed (Participants) | 14 | 12
unitless | -0.9 (1.7) | -1.5 (3.3)

3. Secondary Outcome: Change in Controlled Attenuation Parameter (CAP) Score
Description: The effect of Intermittent fasting on body composition was evaluated using Controlled Attenuation Parameter (CAP) score from Fibroscan. Measurement of controlled attenuation parameter (CAP) is a non-invasive quantitative and qualitative assessment of liver steatosis. CAP measures ultrasonic attenuation (in dB/m) at a frequency of 3.5 MHz (on a go-and-return path). Values range from 100 to 400 dB/m. Higher levels indicate increased hepatic fat.
Time Frame: Assessed before 12-week intervention (baseline) and at week 12
Population: Analysis only includes subjects who completed study through week 12. Unable to obtain a Fibroscan on 10 participants because of body habitus.
Measure: Mean (Standard Deviation); unit: dB/m
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Number analyzed (Participants) | 12 | 7
dB/m | -3.8 (28.3) | -6.6 (74.6)

4. Secondary Outcome: Change in Visceral Adipose Tissue
Description: The effect of intermittent fasting was evaluated by change in visceral adiposity using total body dual energy x-ray absorptiometry (DEXA) between baseline and at week 12.
Time Frame: Assessed before 12-week intervention (baseline) and at week 12
Population: Analysis only includes subjects who completed study through week 12. Ten participants were unable to complete this exam
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Number analyzed (Participants) | 9 | 10
mg | -224 (206) | -149 (541)

5. Secondary Outcome: Change in Lipid Panel Levels
Description: The effect of Intermittent fasting was measured by change in lipid profile levels between baseline and week 12. Lipid profile levels assessed include serum triglyceride, HDL cholesterol, LDL cholesterol, and total cholesterol levels.
Time Frame: Assessed before 12-week intervention (baseline) and at week 12
Population: Analysis only includes subjects who completed study through week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Number analyzed (Participants) | 14 | 14
mg/dL
  Triglyceride | -4.8 (23.5) | 0 (22.9)
  HDL Cholesterol | -1.3 (3.4) | -2.7 (5.7)
  LDL Cholesterol | 1.6 (17.0) | 1.6 (10.9)
  Total Cholesterol | -0.6 (17.4) | -1 (12.5)

6. Secondary Outcome: Change in C-reactive Protein (CRP) Levels
Description: The effect of Intermittent fasting on biomarker of inflammation was measured by C-reactive protein (CRP) levels between baseline and week 12
Time Frame: Assessed before 12-week intervention (baseline) and at week 12
Population: Analysis only includes subjects who completed study through week 12
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Number analyzed (Participants) | 14 | 14
mg/L | 1.7 (4.8) | 0.3 (4.9)

7. Secondary Outcome: Change in Beck Depression Inventory (BDI) Score
Description: The effect of Intermittent fasting on mood was evaluated by change in the Beck Depression Inventory (BDI) score between baseline and week 12. The Beck Depression Inventory (BDI) is a 21-item measure of depression with each question on a 4-point scale ranging from 0=minimal to 3 = more severe (full list score values = 0,1,2,3). Total scores are a sum of individual items. Minimal depression = 0-13, mild depression = 14-19, moderate depression = 20-28, and severe depression = 29-63. The maximum score is 63 and the minimum possible score is zero.
Time Frame: Assessed before 12-week intervention (baseline) and at week 12
Population: Analysis only included subjects who completed study through week 12 and completed the questionnaire
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Number analyzed (Participants) | 5 | 6
Units on a scale | 3.5 (6.8) | 8.6 (7.7)

8. Secondary Outcome: Self-reported Compliance Rate With Assigned Diet
Description: Compliance with assigned diet was assessed by participant self-reported rating. Participants used a self rating score of 0-100% with 0% = noncompliant and 100% = completely compliant with assigned diet. Compliance rate per participant was calculated using average of all daily reported scores. The overall compliance rate was averaged over all participants to get the mean compliance.
Time Frame: Compliance reported at Week 12
Population: Analysis only included subjects who completed study through week 12. 11 subjects did not report their compliance rate.
Measure: Mean (Standard Deviation); unit: Percentage of Compliance
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
Number analyzed (Participants) | 7 | 11
Percentage of Compliance | 80 (16) | 67 (22)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Intermittent Fasting Diet | Standard of Care Diet
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 9/14 | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermittent Fasting Diet (N=14) | Standard of Care Diet (N=16)
Localised oedema (Cardiac disorders) | 1 | 0
Diabetes mellitus (Endocrine disorders) | 2 | 0
Impaired fasting glucose (Endocrine disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 1
Blood bicarbonate decreased (Investigations) | 2 | 1
Blood cholesterol increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 3
Blood glucose increased (Investigations) | 0 | 1
Low density lipoprotein increased (Investigations) | 1 | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the COVID 19 pandemic, study enrollment was stopped and the study did not sufficiently enroll to perform statistical comparisons as originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03489109/Prot_SAP_000.pdf